CLINICAL TRIAL: NCT03805997
Title: Does a Diet With the Recommended Amount of Polyunsaturated Fatty Acids, Increase Their Proportion in Maternal Milk? A Prospective Randomized Open Study
Brief Title: Does a Diet With the Recommended Amount of Polyunsaturated Fatty Acids, Increase Their Proportion in Maternal Milk?
Acronym: ALLAITEMENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC17_8820
Record Dates: First submitted 2019-01-11; First posted 2019-01-16 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding | interventions — Nutrition Assessment; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): consumption of Bleu-Blanc-Cœur products from the 29th week of amenorrhea to the 45th postpartum day
  Interventions: Device: Dietary advice; Other: Consumption of Bleu-Blanc-Coeur products; Biological: Blood sample; Other: Contact; Other: food questionnaire; Other: newborn faeces sample; Other: breast milk sample
- Control Group (Placebo Comparator): no consumption of Bleu-Blanc-Cœur products from the 29th week of amenorrhea to the 45th postpartum day. This group will receive Système U vouchers.
  Interventions: Device: Dietary advice; Other: No consumption of Bleu-Blanc-Coeur products; Biological: Blood sample; Other: food questionnaire; Other: newborn faeces sample; Other: breast milk sample

INTERVENTIONS:
Device: Dietary advice — participants will benefit of dietary device 30-minute dietary advice carried out by a doctor at the University Hospital of Rennes, in order to provide nutritional advice adapted to pregnant women.
Other: Consumption of Bleu-Blanc-Coeur products — consumption of Bleu-Blanc-Cœur products from the 29th week of amenorrhea to the 45th postpartum day
  Arms: Experimental Group
Other: No consumption of Bleu-Blanc-Coeur products — no consumption of Bleu-Blanc-Cœur products from the 29th week of amenorrhea to the 45th postpartum day. This group will receive Système U vouchers.
  Arms: Control Group
Biological: Blood sample — the fatty acid profile of the women red blood cells of the woman wil be test at the inclusion and at 21 days post-partum
Other: Contact — Participants of the group A will be contacted by phone,sms, mail by a technician every 15 days from 7th month of pregnancy to the 8th month of pregnancy and then every week from the 9th month of pregnancy to the 45th postpartum day (except the week of childbirth), in order to collect their consumption data of the delivered food products.
  Arms: Experimental Group
Other: food questionnaire — Participants will have to complete a food questionnaire at the inclusion and at 21 days post-partum
Other: newborn faeces sample — Newborn faeces sample will be collected at 21 Days post partum
Other: breast milk sample — Breast milk sample will be collected at 21 days and 45 days post partum

SUMMARY:
During pregnancy and lactation, the consumption of PUFA n-3, through the consumption of food products that contain more ALA than conventional products, could impact nutritional and non-nutritional breast milk quality (immune criteria, metabolites, hormones), and also the implantation of the intestinal microbiota of the newborn, which is involved in preservation of short term and long term health of the child.

ELIGIBILITY:
Inclusion Criteria:

* women over 18;
* ≤ 28th week of amenorrhea
* having a project of exclusive breastfeeding until at least the 45th day postpartum;
* BMI before pregnancy between 18.5 and 30.0;
* consuming frequently dairy products, eggs, meat (pork, beef, poultry);
* accepting the consumption of all food products delivered;
* written consent received and signed.

Non-inclusion criteria:

* multiple pregnancy;
* eating disorders or suspicion (defined by SCOFF score);
* vegetarian, vegan or flexitarian;
* allergic to food product(s) involved in the study;
* home with more than 2 adults and 3 children (excluding foetus);
* adults on legal protection (guardianship, trusteeship…), persons deprived of liberty;

Exclusion Criteria:

* Interruption of breastfeeding before the 21st postpartum day
* Prematurity: childbirth before the 37th week of amenorrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Level of α-linolenic acid in milk | on the 21st postpartum day.
  The primary evaluation criterion is the level of α-linolenic acid in milk on the 21st postpartum day.

SECONDARY OUTCOMES:
The α-linolenic acid level of breast milk | at the 45th postpartum day;
  The α-linolenic acid level of breast milk at the 45th postpartum day;
The fatty acid content of breast milk ; | on the 21st and the 45th postpartum days
  The fatty acid content of breast milk on the 21st and the 45th postpartum days;
The cytokine content of breast milk | on the 21st and the 45th postpartum days
  The cytokine content of breast milk on the 21st and the 45th postpartum days: IL-6, TNFα, TGFβ
The immunoglobulin A and G content of breast milk | on the 21st and the 45th postpartum days;
  The immunoglobulin A and G content of breast milk on the 21st and the 45th postpartum days;
The lactoferrin content (antimicrobial factor) of breast milk | on the 21st and the 45th postpartum days;
  The lactoferrin content (antimicrobial factor) of breast milk on the 21st and the 45th postpartum days;
The hormone content of breast milk | on the 21st and the 45th postpartum days
  The hormone content of breast milk on the 21st and the 45th postpartum days: adiponectin, leptin, insulin;
The oligosaccharide content of breast milk | on the 21st and the 45th postpartum days
  The oligosaccharide content of breast milk on the 21st and the 45th postpartum days;
The breast milk microbiota content | on the 21st and the 45th postpartum days
  The breast milk microbiota content on the 21st and the 45th postpartum days;
the bacterial intestinal microbiota content from the feces of the newborn | on the 21st postpartum day;
  the bacterial intestinal microbiota content from the feces of the newborn on the 21st postpartum day;
Fatty acid content | before the 7th month of pregnancy and on the 21st postpartum day.
  the fatty acid content of the women red blood cells of the woman before the 7th month of pregnancy and on the 21st postpartum day.
The breast milk lipidome | on the 21st postpartum day
  the breast milk lipidome on the 21st postpartum day: 26 lipid classes comprising more than 300 different lipid species (in addition to the total fatty acid analyses of breast milk, in order to make a complete description of the lipid species provided);
The maternal milk metabolome | On the 21st postpartum day
  the maternal milk metabolome on the 21st postpartum day: metabolites, hormones and other signal molecules (this analysis complements the previous ones by producing a complete description of non-lipid metabolites in breast milk);

CONTACTS AND LOCATIONS:
Locations (1):
- CIC CHU de Rennes, Rennes, France